CLINICAL TRIAL: NCT06279130
Title: Pan-tumor Neoadjuvant Basket Study of Immune Check-point Inhibition and Novel Immuno-oncology Combinations
Acronym: NEOASIS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N23NEO
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Resectable MMR-deficient Solid Tumors; Resectable MMR-proficient Solid Tumors
MeSH Terms: interventions — balstilimab

STUDY DESIGN:
Intervention Model Description: Basket, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- pMMR Safety run-in 1 (Experimental): 5 Patients will be included and will be treated with 2 cycles of neoadjuvant immunotherapy consisting of 450mg balstilimab and 25mg botensilimab in Cycle 1 and 450mg balstilimab in Cycle 2 followed by surgery
  Interventions: Drug: botensilimab; Drug: balstilimab
- pMMR Safety run-in 2 (Experimental): 5 Patients will be included and will be treated with 2 cycles of neoadjuvant immunotherapy consisting of 450mg balstilimab and 50mg botensilimab in Cycle 1 and 450mg balstilimab in Cycle 2 followed by surgery
  Interventions: Drug: botensilimab; Drug: balstilimab
- dMMR Safety run-in 1 (Experimental): 5 Patients will be included and will be treated with 2 cycles of neoadjuvant immunotherapy consisting of 450mg balstilimab and 25mg botensilimab in Cycle 1 and 450mg balstilimab in Cycle 2 followed by surgery
  Interventions: Drug: botensilimab; Drug: balstilimab
- dMMR Safety run-in 2 (Experimental): 5 Patients will be included and will be treated with 2 cycles of neoadjuvant immunotherapy consisting of 450mg balstilimab and 50mg botensilimab in Cycle 1 and 450mg balstilimab in Cycle 2 followed by surgery
  Interventions: Drug: botensilimab; Drug: balstilimab
- dMMR Colorectal basket (Experimental): Patients with resectable colon and rectal cancer will be treated with the regimen assesses as safe and feasible in the dMMR safety run-in. Treatment will be administered at day 1 and day 22 followed by surgery 8 weeks after registration. Accrual will be temporarily halted after accrual of the first 8 patients. If >2 major pathological responses are observed accrual will continue to a total of 18 patients.
  Interventions: Drug: botensilimab; Drug: balstilimab
- dMMR Gynaecological oncology basket (Experimental): Patients with resectable endometrial, cervical and ovarian cancer will be treated with the regimen assessed as safe and feasible in the dMMR safety run-in. Treatment will be administered at day 1 and day 22 followed by surgery 8 weeks after registration. Accrual will be temporarily halted after accrual of the first 8 patients. If >2 major pathological responses are observed accrual will continue to a total of 18 patients.
  Interventions: Drug: botensilimab; Drug: balstilimab
- dMMR Upper gastro-intestinal cancer basket (Experimental): Patients with resectable oesophageal (adenocarcinoma), gastro-oesophageal junction, gastric and small bowel cancer will be treated with the regimen assessed as safe and feasible in the dMMR safety run-in. Treatment will be administered at day 1 and day 22 followed by surgery 8 weeks after registration. Accrual will be temporarily halted after accrual of the first 8 patients. If >2 major pathological responses are observed accrual will continue to a total of 18 patients.
  Interventions: Drug: botensilimab; Drug: balstilimab
- dMMR "other cancers" baskets (Experimental): Patients with resectable solid tumors of various origins such as but not limited to breast-, prostate-, bladder cancer, Head&Neck SCC, oesophageal SCC and sarcoma will be treated with the regimen assessed as safe and feasible in the dMMR safety run-in. Treatment will be administered at day 1 and day 22 followed by surgery 8 weeks after registration. Accrual will be temporarily halted after accrual of the first 8 patients. If >2 major pathological responses are observed accrual will continue to a total of 18 patients.
  Interventions: Drug: botensilimab; Drug: balstilimab

INTERVENTIONS:
Drug: botensilimab — Anti cytotoxic T-lymphocyte associated protein-4 (anti-CTLA4)
Drug: balstilimab — Anti programmed cell death protein-1 (anti-PD1)

SUMMARY:
In this study, the efficacy of botensilimab and balstilimab in mismatch repair deficient (dMMR) and mismatch repair proficient (pMMR) tumors will be assessed.

DETAILED DESCRIPTION:
The NEOASIS study is an adaptive, pan-cancer, single-center, open-label, basket study assessing the efficacy of botensilimab and balstilimab in patients with resectable dMMR and pMMR solid tumors of various origins. Patients will be included in baskets according to tumor type and mismatch repair (MMR) status and will receive 2 cycles of immunotherapy followed by surgery.

The trial will commence with two safety run-in cohorts: one for patients with dMMR tumors and one for patients with pMMR tumors that will run in parallel. These safety run-in cohort will be used to assess safety and feasibility of pre-operative botensilimab + balstilimab. Data from the safety run-in cohorts will be used to determine the dosing and scheduling to be used in the MMR-specific cohorts of the main study. Safety will be assessed according to dose limiting toxicities. In the run-in cohorts, the first five patients will receive botensilimab 25mg intravenously (IV) on Day1 plus balstilimab 450mg IV on Day1 and Day22. Patients 6-10 will receive botensilimab 50mg IV on Day1 plus balstilimab 450mg IV on Day1 and Day22 followed by surgery 8 weeks after registration.

After full accrual of the run-in cohorts, MMR-specific baskets including a "other cancers" basket will start accrual with the optimal dose and schedule as determined in the safety run-in followed by surgery 8 weeks after registration. The MMR-specific baskets are designed with a Simon's 2 stage design in which first 8 patients will be included, if in the first 8 patients >2 Major pathological responses are reported (defined as ≤10% residual viable tumor) accrual of 10 more patients will continue for a total of 18 patients per basket.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Patients at least 18 years of age
3. Non-metastatic, newly diagnosed dMMR and pMMR cancers either fitting within a specific basket or in the "other" cohort (e.g. sarcoma, head and neck cancers, anal cancer, esophageal SCC)
4. In case of pMMR tumors: no indication for neoadjuvant therapy according to standard of care, unless adjuvant treatment is considered a standard of care alternative;
5. Eligible for study biopsy
6. World health organization (WHO) performance status of 0 or 1
7. Screening laboratory tests must meet the following criteria and should be obtained within 7 days prior to randomization/registration: White blood cell count (WBC > 2.0 x 10^9/L, Absolute neutrophil count (ANC) > 1.5x10^9/L, platelets > 100 x 10^9/L, Hemoglobin > 5.0mmol/L. Transfusion is allowed to obtain an adequate hemoglobin level. Liver function tests: total bilirubin < 1.5 upper limit of normal (ULN) (except for subjects with Gilbert syndrome, who can have total bilirubin <3.0 mg/dL); alkaline phosphatase <1.5 ULN; transaminases (ASAT/ALAT) <3 x ULN; Lactate dehydrogenase (LDH) < 1.5x ULN; Creatinine clearance (Cockcroft-Gault) of >45 ml/min, Albumin > 3.0 g/dL
8. Women of childbearing potential (WOCBP)* must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 20 weeks after the last dose of investigational drug, Non-childbearing potential is defined as:

   1. Postmenopausal: ≥ 50 years of age and has not had menses for greater than 1 year.
   2. Amenorrheic for ≥ 2 years without a hysterectomy and bilateral oophorectomy and a follicle- stimulating hormone value in the postmenopausal range upon pre-study(screening) evaluation.
   3. Status is post-hysterectomy, bilateral oophorectomy, or tubal ligation.
9. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of cycle 1 day 1
10. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving the study treatment and who are sexually active with WOCBP (excluding azoospermic men) will be instructed to adhere to contraception for a period of 28 weeks after the last dose of investigational drug and are not allowed to donate sperm during that timeframe.

Exclusion Criteria:

1. Signs of distant metastases on imaging and physical examination
2. Clinical obstruction
3. Clinical symptoms or radiological suspicion of perforation
4. Previous treatment with immune checkpoint inhibitors including but not limited to anti-CTLA4 or anti-PD1
5. Prior chemotherapy for any cancer
6. Radiotherapy prior to or planned post-surgery radiotherapy for disease under study
7. Active malignancies other than disease under study within 3 years prior to inclusion, except for malignancies with a negligible recurrence rate (e.g. <10% in 5 years)
8. Allergies and Adverse Drug Reaction:

   1. History of allergy to study drug components
   2. History of severe hypersensitivity reaction to any monoclonal antibody
9. Intercurrent illnesses, including but not limited to infections, unstable angina pectoris
10. Underlying medical conditions that, in the investigator's opinion, will make the administration of the study drug hazardous or obscure the interpretation of toxicity determination of adverse events
11. Positive test for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
12. History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
13. Active autoimmune disease or a documented history of autoimmune disease, or other medical conditions requiring systemic steroid or immunosuppressive medications, except for subjects with vitiligo, diabetes mellitus type 1, hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis or resolved childhood asthma/atopy not requiring systemic treatment
14. Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
15. Live vaccines in the 4 weeks prior to inclusion
16. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
17. Current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2029-01-29 (Estimated); Study Completion 2034-01-29 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate | Week 8
  Percentage of patients in which a major pathologic response (MPR) is reported, defined as <10% residual viable tumor (RVT) in the resection specimen.

SECONDARY OUTCOMES:
Pathological response rates | Week 8
  Pathologic complete response (pCR) defined as no RVT in the primary tumor and locoregional lymph nodes; partial pathologic response (≤50% RVT) and no pathologic response (>50% RVT)
Event free survival | 3 years
  Event-free survival defined as time from registration to the date of disease progression, local, regional or distant recurrence, occurrence of a second primary cancer or death from any cause.
Disease free survival | 3 years
  Disease free survival defined as the time from surgery to disease recurrence during follow-up which consists of either local or regional recurrence, metastatic disease or disease-related death.
Overall survival | 5 years
  Overall survival defined as time from registration until death from any cause.
Radiological response | Week 8
  Radiological response measured according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Chalabi, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No